CLINICAL TRIAL: NCT06898216
Title: Flexible Ureteroscopy With Steerable Versus Conventional Flexible and Navigable Suction Ureteral Access Sheath (FANS) Utility in Less Than 2cm Lower Pole Stones Treatment: a Multicenter, Randomized Superiority Trial (SCULPT Trial)
Brief Title: Steerable vs Conventional FANS for <2cm Lower Pole Stone Treatment: SCULPT Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: the third Medical Center, PLA General Hospital (Unknown); First Affiliated Hospital of Chongqing Medical University (Other); Peking University People's Hospital (Other); The Second Affiliated Hospital of Kunming Medical University (Other); The Fifth Affiliated Hospital, Sun Yat-sen University (Unknown); Henan Provincial People's Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Wuhan Hospital of Traditional Chinese Medicine (Other); Dongguan People's Hospital (Other Government); Changzhou No.2 People's Hospital (Other); Dongguan Tungwah Hospital (Other); Panzhihua Central Hospital (Other); Yan'an Hospital of Kunming City (Unknown); NO.1 People's Hospital of Dali City (Unknown); Huadu District People's Hospital of Guangzhou (Other); Jiangmen Central Hospital (Other); Shaoyang Central Hospital (Unknown); Guangzhou Medical University Affiliated Qingyuan Hospital (Unknown); Dongguan Kanghua Hospital (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ES-2025-033
Record Dates: First submitted 2025-03-16; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Kidney Stones
Keywords: flexible ureteroscopy; flexible and navigable suction ureteral access sheath; FANS; lower pole; renal stones
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steerable FANS Arm (Experimental): Participants assigned to this arm will undergo flexible ureteroscopy using the novel steerable flexible and navigable suction ureteral access sheath (FANS). This device incorporates an active deflection mechanism that allows for independent adjustment to optimize navigation into the lower pole calyx. The procedure is performed under general anesthesia with a standardized 7.5 Fr digital flexible ureteroscope, using a 200 µm holmium laser (energy settings ≤30 W) for lithotripsy, and continuous negative-pressure suction for stone fragment aspiration. Adjunct devices (e.g., stone baskets) may be utilized if necessary.
  Interventions: Device: Steerable FANS
- Conventional FANS Arm (Active Comparator): Participants assigned to this arm will receive flexible ureteroscopy using the conventional flexible and navigable suction ureteral access sheath (FANS), which relies on passive deflection provided by the ureteroscope for navigation into the lower pole calyx. The procedure is conducted under general anesthesia with a 7.5 Fr digital flexible ureteroscope, employing a 200 µm holmium laser (energy settings ≤30 W) for lithotripsy and continuous negative-pressure suction for fragment removal. Adjunctive retrieval tools (e.g., stone baskets) may be used as required.
  Interventions: Device: Conventional FANS

INTERVENTIONS:
Device: Steerable FANS — This device is designed for flexible ureteroscopy procedures in patients with lower pole renal stones ≤2 cm. It features an active deflection mechanism that enables independent adjustment to enhance access into the lower pole calyx. The description focuses solely on the device and does not include procedural details already provided in the arm description.
  Other Names: Steerable Flexible and Navigable Suction Ureteral Access Sheath
  Arms: Steerable FANS Arm
Device: Conventional FANS — This device is intended for use in flexible ureteroscopy for lower pole renal stone management. It relies on passive deflection provided by the flexible ureteroscope for navigation into the lower pole calyx. The description is limited to the device characteristics without duplicating procedural details from the arm description.
  Other Names: Conventional Flexible and Navigable Suction Ureteral Access Sheath
  Arms: Conventional FANS Arm

SUMMARY:
This multicenter, randomized, controlled superiority trial (the SCULPT trial) aims to compare the efficacy and safety of a novel steerable flexible and navigable suction ureteral access sheath (FANS) versus the conventional FANS in the treatment of lower pole renal stones ≤2 cm. Lower pole stones are particularly challenging due to the narrow infundibular-pelvic anatomy that limits the maneuverability of standard FANS. The steerable FANS incorporates an active deflection mechanism that allows for independent control, potentially improving the success rate of accessing the lower pole calyx, performing laser lithotripsy, and aspirating stone fragments without additional adjuncts.

A total of 400 patients from 20 high-volume urological centers in China (approximately 20 patients per center) will be randomized in a 1:1 ratio to receive either steerable FANS or conventional FANS during flexible ureteroscopy. Primary outcome measures include the success rate of FANS navigation into the lower pole calyx as evidenced by direct stone visualization, effective laser lithotripsy, and successful stone aspiration. Secondary outcomes will assess immediate and 1-month stone-free rates, operative time, complication rates, instrument durability, and improvements in quality of life. This study is expected to provide critical evidence to guide clinical decision-making and potentially improve treatment efficiency for challenging lower pole renal stones.

DETAILED DESCRIPTION:
This trial is designed in response to the current challenges faced in the management of lower pole renal stones using flexible ureteroscopy, particularly when using conventional FANS. The narrow calyceal angles and complex lower pole anatomy can impede the passage of the access sheath, thereby limiting the efficiency of stone fragmentation and clearance. The innovative steerable FANS overcomes these limitations by offering an independent, active deflection mechanism that facilitates a greater range of movement, thus optimizing the access to lower pole calyces.

Background and Objectives Lower pole stones are notoriously difficult to treat due to their anatomical position and the limited maneuverability of conventional ureteral access sheaths. The new steerable FANS, with its deflection lever at the distal handle, allows for active, independent adjustment under endoscopic guidance, which may result in a higher success rate of reaching the lower pole and more efficient stone clearance. The primary objective of this trial is to compare the success rate of FANS navigation into the lower pole renal calyx between the steerable and conventional devices. Secondary objectives include the evaluation of immediate (within 24 hours) and 1-month stone-free rates, operative time, length of hospital stay, usage of auxiliary devices (e.g., stone baskets), instrument damage rates, complication rates (graded by the Clavien-Dindo system), and the impact on patient quality of life (assessed via the Wisconsin Stone QoL questionnaire).

Study Design and Methods

Trial Type:

This is a multicenter, prospective, single-blind, superiority, randomized controlled trial.

Study Setting and Participants:

The study will be conducted at 20 high-volume urological centers across China, with each center recruiting approximately 20 patients. Eligible participants are adults aged 18-75 years, diagnosed with a single lower pole renal stone ≤2 cm (confirmed by CT) and who meet all inclusion and exclusion criteria.

Randomization and Group Allocation:

A centralized, stratified randomization process (1:1 ratio) will allocate patients to either the steerable FANS or conventional FANS group. Random sequences will be generated electronically using permuted blocks within each center to maintain allocation concealment.

Interventions:

All patients will undergo flexible ureteroscopy under general anesthesia with standardized use of 7.5 Fr digital flexible ureteroscopes. Preoperative imaging (contrast-enhanced CT urography) will assess stone size, location, and anatomical parameters. Depending on ureteral diameter, an appropriate FANS (either 11/13 Fr or a smaller version) will be selected. Laser lithotripsy will be performed using a 200 µm laser fiber (energy settings ≤30 W) alongside continuous negative-pressure suction to aspirate stone fragments. If the sheath cannot be navigated into the lower pole due to anatomical constraints, an adjunct stone basket may be employed.

Outcome Measures:

Primary Outcome:

The success rate of FANS navigation into the lower pole calyx, defined as the sheath reaching the calyx, performing effective laser lithotripsy, and aspirating stone fragments without additional adjuncts.

Secondary Outcomes:

These include the immediate (24-hour) and final (1-month) stone-free rates (defined as no residual stone or fragments >2 mm on CT), operative time, duration of hospital stay, intraoperative usage of adjunct devices, damage rates of the ureteroscope and FANS, complications within one month (graded by Clavien-Dindo), and quality of life improvements as measured by the Wisconsin Stone QoL questionnaire.

Follow-up and Data Collection:

Patients will undergo a low-dose CT scan within 24 hours postoperatively to assess the immediate stone-free status, with a follow-up CT at 1 month for final assessment. Clinical data, including operative details and follow-up results, will be recorded in standardized case report forms (CRFs) at each center. This will ensure consistency and completeness of data across the multicenter trial.

Sample Size and Statistical Analysis:

Based on preliminary data showing a 60% success rate with conventional FANS and an anticipated 80% with the steerable FANS, with a superiority margin of 6%, a total of 400 participants (200 per group) has been calculated to achieve 80% power at a one-sided α of 2.5%, accounting for potential dropouts. Statistical analyses will be conducted using SPSS software, with continuous variables analyzed via t-tests or Mann-Whitney U tests (depending on data distribution) and categorical variables assessed using chi-square or Fisher's exact tests. Multivariate analyses will be performed where necessary, and results will be presented with 95% confidence intervals.

Quality Control and Safety Monitoring:

All participating centers will undergo standardized training to ensure uniformity in surgical procedures and data collection. Monthly monitoring visits will verify protocol adherence and data integrity. Any adverse events will be meticulously recorded and reported promptly to the Ethics Committee, with regular cumulative safety reviews performed by the principal investigator.

Significance and Expected Outcomes This trial is the first head-to-head comparison of steerable versus conventional FANS in the management of lower pole renal stones. If the steerable FANS demonstrates superiority in navigating the lower pole and enhancing stone clearance efficiency, it could transform the current endourological approach to challenging renal calculi. In addition, the comprehensive evaluation of instrument durability and complication profiles will aid in economic assessments and inform patient counseling regarding procedural risks and benefits. Ultimately, the findings of this study are expected to contribute robust evidence toward optimizing clinical strategies, improving patient outcomes, and potentially expanding the indications for flexible ureteroscopy in complex renal stone management.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 years
* Diagnosed with a single lower pole renal stone ≤2 cm by CT
* American Society of Anesthesiology (ASA) score of 1-3
* Ability to provide written informed consent
* Willingness and ability to comply with trial procedures and follow-up

Exclusion Criteria:

* Patients with urinary tract anatomical abnormalities (e.g., horseshoe kidney, ileal conduit)
* Untreated urinary tract infection
* Presence of multiple stones or stones located outside the lower pole
* Absolute contraindications to flexible ureteroscopy
* Inability to understand or complete trial documentation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-03-16 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Success Rate of Lower Pole Navigation | Periprocedural (Day of Procedure)
  This outcome is defined as the proportion of cases in which the FANS (either steerable or conventional) successfully navigates into the lower pole renal calyx. Success is evidenced by the ability to directly visualize the stone, perform effective laser lithotripsy, and aspirate stone fragments without requiring additional adjunctive devices.

SECONDARY OUTCOMES:
Immediate Stone-Free Rate | Day 1
  Proportion of patients with no residual stones or fragments >2 mm on CT scan performed within 24 hours postoperatively.
Final Stone-Free Rate | 1 month
  Proportion of patients with complete stone clearance or fragments ≤2 mm, as confirmed by low-dose CT scan at 1 month postoperatively.
Operative Time | Periprocedural (Day of Procedure)
  Duration from the insertion of the flexible ureteroscope into the urethra until the completion of double-J stent placement.
Duration of Hospital Stay | Periprocedural (Day of Procedure through Discharge)
  Total number of whole days from the day of surgery to the day of discharge.
Use of Adjunct Devices | Recorded during the procedure
  Frequency of intraoperative usage of additional retrieval tools (e.g., stone baskets) when the FANS is unable to reach the lower pole.
Instrument Damage Rates | Periprocedural (Day of Procedure)
  Incidence of intraoperative damage to the flexible ureteroscope and FANS requiring repair or replacement.
Complication Rate | Up to 1 month
  Incidence and severity of complications occurring up to 1 month post-procedure, graded according to the Clavien-Dindo classification system.
Quality of Life Improvement | Baseline and 1 month
  Changes in patient-reported quality of life as assessed by the Wisconsin Stone Quality of Life (WISQOL) questionnaire. The questionnaire is scored on a scale from 0 to 100, where higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, M.D., Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Urology, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuen SKK Steffi, Liu S, Gauhar V, Mai H, He W, Hu H, Ke C, Dai Y, Shan L, Jiang Y, Yuan J, Cao Z, Zuo L, Yang C, Bai B, Bi X, Zhao H, Xi M, Ding N, Deng S, Tang S, Zeng J, Du J, Wu W, Ma J, Zhong W, Zhao Z, Liu Y, de la Rosette J, Zeng G, Zhu W. Steerable versus Conventional flexible and navigable suction ureteral access sheath (FANS) flexible Ureteroscopy for Lower Pole stones Treatment: study protocol for a multicentre, randomised superiority trial (SCULPT trial). BMJ Open. 2025 Dec 2;15(12):e103866. doi: 10.1136/bmjopen-2025-103866. PMID 41338650